CLINICAL TRIAL: NCT04735211
Title: Risk Factors to Develop Chronic Postsurgical Pediatric Pain: An Observational Study
Brief Title: Chronic Postsurgical Pediatric Pain. Evaluation Risk Factors to Develop Chronic Postsurgical Pain in Children and Adolescents Undergoing Surgery in a First Level Hospital
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Guillermo Ceniza Bordallo (Other)
Responsible Party: Sponsor-Investigator, Guillermo Ceniza Bordallo, Principal Investigator, Universidad Complutense de Madrid
Organization: Universidad Complutense de Madrid (Other)
Other Study IDs: 20/618
Record Dates: First submitted 2021-01-12; First posted 2021-02-03 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Chronic Postoperative Pain; Pediatric ALL
Keywords: Chronic Postsurgical Pediatric Pain
MeSH Terms: conditions — Pain, Postoperative; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children whom develop chronic postsurgical pain: Children whom had chronic pain at 3 moths after surgery
  Interventions: Procedure: Surgery
- Children whom not develop chronic postsurgical pain: Children whom not develop chronic pain at 3 moths after surgery

INTERVENTIONS:
Procedure: Surgery — Pediatric Surgery with hospitalized
  Groups: Children whom develop chronic postsurgical pain

SUMMARY:
Chronic postsurgical pain had number of prevalence on 20%. Its derivates from risk factors, but recent research provide new potential risk factors to develop chronic postsurgical pediatric pain.

To increase the body of knowledge, an observational study is proposed in pediatric patients undergoing surgical intervention.

DETAILED DESCRIPTION:
A cohort of pediatric patients undergoing surgery will be followed at the Maternal and Child Hospital October 12, Madrid. The group of patients that develops post-surgical chronic pain and the group that does not develop it will be observed, and risk factors will be studied.

Before the surgical intervention, the risk factors described in the literature will be analyzed. Children will be followed up to 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children with age from 4 years to 18 years. Undergoing surgery for any surgical specialty. ASA Status (American Society of Anesthesiologist) from I to III.

Exclusion Criteria:

* Children who do not understand and speak Spanish correctly. Children with verbal communication problems.

Ages: 4 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric Population undergoing surgical intervention.
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Type of surgery | 1 day presurgery
  Surgery Specialty.
Previous pathologies | 1 day presurgery
  Previous pathologies
Baseline Child Catastrophizing | 1 day presurgery
  Assess by Child Catastrophizing scale.The Pain Catastrophizing Scale-Child (PCS-C);is a validated self-report measure that is used to assess negative thinking associated with pain. The PCS-C include 13 items, which are rated on a 5-point scale ranging from 0 = "not at all true" to 4 = "very true." The items are divided across three subscales: rumination (4 items, e.g. "When I have pain, I can't keep it out of my mind"), magnification (3 items, e.g. "When I have pain, I keep thinking of other painful events") and helplessness (6 items, e.g. "When I have pain, I feel like I can't go on"
Change of Child Catastrophizing at 3 moths postsurgery | 3 months
  Assess by Child Catastrophizing scale.The Pain Catastrophizing Scale-Child (PCS-C);is a validated self-report measure that is used to assess negative thinking associated with pain. The PCS-C include 13 items, which are rated on a 5-point scale ranging from 0 = "not at all true" to 4 = "very true." The items are divided across three subscales: rumination (4 items, e.g. "When I have pain, I can't keep it out of my mind"), magnification (3 items, e.g. "When I have pain, I keep thinking of other painful events") and helplessness (6 items, e.g. "When I have pain, I feel like I can't go on"
Change of Child Catastrophizing at 6 moths postsurgery | 6 months
  Assess by Child Catastrophizing scale.The Pain Catastrophizing Scale-Child (PCS-C);is a validated self-report measure that is used to assess negative thinking associated with pain. The PCS-C include 13 items, which are rated on a 5-point scale ranging from 0 = "not at all true" to 4 = "very true." The items are divided across three subscales: rumination (4 items, e.g. "When I have pain, I can't keep it out of my mind"), magnification (3 items, e.g. "When I have pain, I keep thinking of other painful events") and helplessness (6 items, e.g. "When I have pain, I feel like I can't go on"
Baseline Child Anxiety | 1 day presurgery
  Assess by Child Anxiety Symptoms Scale (CPASS) is a 20-item scale for children adapted from the adult PASS-20. For each statement, children are asked to rate the extent to which they think, act, or feel that way on a scale from 0 (''never think, act or feel that way'') to 5 (''always think, act, or feel that way''). Total scores range from 0 to 100, with higher scores indicating higher levels of pain anxiety.
Change of Child Anxiety at 3 moths postsurgery | 3 moths
  Assess by Child Anxiety Symptoms Scale (CPASS) is a 20-item scale for children adapted from the adult PASS-20. For each statement, children are asked to rate the extent to which they think, act, or feel that way on a scale from 0 (''never think, act or feel that way'') to 5 (''always think, act, or feel that way''). Total scores range from 0 to 100, with higher scores indicating higher levels of pain anxiety.
Change of Child Anxiety at 6 moths postsurgery | 6 moths
  Assess by Child Anxiety Symptoms Scale (CPASS) is a 20-item scale for children adapted from the adult PASS-20. For each statement, children are asked to rate the extent to which they think, act, or feel that way on a scale from 0 (''never think, act or feel that way'') to 5 (''always think, act, or feel that way''). Total scores range from 0 to 100, with higher scores indicating higher levels of pain anxiety.
Baseline Pain Interference | 1 day presurgery
  Asess by PROMIS-Pediatric Pain Interference Scale (PPIS): The 8-item PPIS assesses how the child's pain has interfered with certain aspects of their life over the past 7 days (eg, sleep, attention, schoolwork, physical activities, emotion). Each item is rated on a 5-point scale ranging from "never" to "almost always". Scores range from 0 to 32 where higher scores indicate greater pain-related functional impairment.
Change of Pain Interference at 3 moths postsurgery | 3 moths
  Asess by PROMIS-Pediatric Pain Interference Scale (PPIS): The 8-item PPIS assesses how the child's pain has interfered with certain aspects of their life over the past 7 days (eg, sleep, attention, schoolwork, physical activities, emotion). Each item is rated on a 5-point scale ranging from "never" to "almost always". Scores range from 0 to 32 where higher scores indicate greater pain-related functional impairment.
Change of Pain Interference at 6 moths postsurgery | 6 moths
  Asess by PROMIS-Pediatric Pain Interference Scale (PPIS): The 8-item PPIS assesses how the child's pain has interfered with certain aspects of their life over the past 7 days (eg, sleep, attention, schoolwork, physical activities, emotion). Each item is rated on a 5-point scale ranging from "never" to "almost always". Scores range from 0 to 32 where higher scores indicate greater pain-related functional impairment.
Baseline Child Fear of pain | 1 day presurgery
  Assess by The Fear of Pain Questionnaire-Children (FOPQ-C): Is a validated self-report measure that used to asses fear of pain in children. The FOPQ-C include 23 ítems, which are rated on a 5-point scale ranging 0=" not at all" 5="very true". The items are divided across two subscales: fear of pain, and avoidance activities.
Change of Child Fear of pain at 3 moths postsurgery | 3 moths
  Assess by The Fear of Pain Questionnaire-Children (FOPQ-C): Is a validated self-report measure that used to asses fear of pain in children. The FOPQ-C include 23 ítems, which are rated on a 5-point scale ranging 0=" not at all" 5="very true". The items are divided across two subscales: fear of pain, and avoidance activities.
Change of Child Fear of pain at 6 moths postsurgery | 6 moths
  Assess by The Fear of Pain Questionnaire-Children (FOPQ-C): Is a validated self-report measure that used to asses fear of pain in children. The FOPQ-C include 23 ítems, which are rated on a 5-point scale ranging 0=" not at all" 5="very true". The items are divided across two subscales: fear of pain, and avoidance activities.
Baseline Child Kinesiophobia | 1 day presurgery
  Assess by The Tampa Scale Kinesiophobia (TSK-11). Is a 11-item scale that measures fear of move- ment-evoked pain and injury. Scale items ranges from 0 (strongly disagree) to 4 (strongly agree) with 4 reversed- scored items. Total scores range from 25 to 56 with higher scores indicative of a greater fear of movement.
Change of Child Kinesiophobia at 3 moths postsurgery | 3 moths
  Assess by The Tampa Scale Kinesiophobia (TSK-11). Is a 11-item scale that measures fear of move- ment-evoked pain and injury. Scale items ranges from 0 (strongly disagree) to 4 (strongly agree) with 4 reversed- scored items. Total scores range from 25 to 56 with higher scores indicative of a greater fear of movement.
Change of Child Kinesiophobia at 6 moths postsurgery | 6 moths
  Assess by The Tampa Scale Kinesiophobia (TSK-11). Is a 11-item scale that measures fear of move- ment-evoked pain and injury. Scale items ranges from 0 (strongly disagree) to 4 (strongly agree) with 4 reversed- scored items. Total scores range from 25 to 56 with higher scores indicative of a greater fear of movement.
Baseline Health-related Quality of Life in Children | 1 day presurgery
  Pediatric Quality of Life version 4.0 (PedsQL 4.0), which is a widely used measure of health-related quality of life in children. The PedsQL consists of 23-items and includes both child-report (for those age 8 and over). The PedsQL assesses the following four domains of functioning: physical, emotional, social, and school and items are rated on a five-point Likert-type scale that ranges from 0 (never a problem) to 4 (almost always a problem). Items are converted to create a 0-100 scale, with higher scores reflecting higher quality of life.
Change of Health-related Quality of Life in Children at 3 moths postsurgery | 3 moths
  Pediatric Quality of Life version 4.0 (PedsQL 4.0), which is a widely used measure of health-related quality of life in children. The PedsQL consists of 23-items and includes both child-report (for those age 8 and over). The PedsQL assesses the following four domains of functioning: physical, emotional, social, and school and items are rated on a five-point Likert-type scale that ranges from 0 (never a problem) to 4 (almost always a problem). Items are converted to create a 0-100 scale, with higher scores reflecting higher quality of life.
Change Health-related Quality of Life in Children at 6 moths postsurgery | 6 moths
  Pediatric Quality of Life version 4.0 (PedsQL 4.0), which is a widely used measure of health-related quality of life in children. The PedsQL consists of 23-items and includes both child-report (for those age 8 and over). The PedsQL assesses the following four domains of functioning: physical, emotional, social, and school and items are rated on a five-point Likert-type scale that ranges from 0 (never a problem) to 4 (almost always a problem). Items are converted to create a 0-100 scale, with higher scores reflecting higher quality of life.
Baseline Pain intensity | 1 day presurgery
  Assess by The Numerical Rating Scale (NRS) is a verbally administered scale that measures pain intensity (''how much pain do you feel right now?''). The NRS can also be used to measure pain unpleas- antness (''how unpleasant/horrible/yucky is the pain right now?''). The end points represent the extremes of the pain experience.
Change of Pain intensity 3 moths postsurgery | 3 moths
  Assess by The Numerical Rating Scale (NRS) is a verbally administered scale that measures pain intensity (''how much pain do you feel right now?''). The NRS can also be used to measure pain unpleas- antness (''how unpleasant/horrible/yucky is the pain right now?''). The end points represent the extremes of the pain experience.
Change of Pain intensity at 6 moths postsurgery | 6 moths
  Assess by The Numerical Rating Scale (NRS) is a verbally administered scale that measures pain intensity (''how much pain do you feel right now?''). The NRS can also be used to measure pain unpleas- antness (''how unpleasant/horrible/yucky is the pain right now?''). The end points represent the extremes of the pain experience.

SECONDARY OUTCOMES:
Baseline Parent Anxiety | 1 day presurgery
  Assess by Pain Anxiety Symptoms Scale-Short Form (PASS-20) PASS-2022 consists of 20 items that measure the fear and anxiety-related thoughts, feelings, behaviors, and physical sensations that accompany the experience and anticipation of pain. Each item is rated on a scale of 0 (never) to 5 (always) and total scores range from 0 to 100. The PASS-20 has four subscales: cognitive, escape/avoidance, fear, and physiological anxiety.
Change of Parent Anxiety at 3 moths postsurgery | 3 moths
  Assess by Pain Anxiety Symptoms Scale-Short Form (PASS-20) PASS-2022 consists of 20 items that measure the fear and anxiety-related thoughts, feelings, behaviors, and physical sensations that accompany the experience and anticipation of pain. Each item is rated on a scale of 0 (never) to 5 (always) and total scores range from 0 to 100. The PASS-20 has four subscales: cognitive, escape/avoidance, fear, and physiological anxiety.
Change of Parent Anxiety at 6 moths postsurgery | 6 moths
  Assess by Pain Anxiety Symptoms Scale-Short Form (PASS-20) PASS-2022 consists of 20 items that measure the fear and anxiety-related thoughts, feelings, behaviors, and physical sensations that accompany the experience and anticipation of pain. Each item is rated on a scale of 0 (never) to 5 (always) and total scores range from 0 to 100. The PASS-20 has four subscales: cognitive, escape/avoidance, fear, and physiological anxiety.
Baseline Parent Catastrophizing | 1 day presurgery
  The Pain Catastrophizing Scale-Parent report (PCS-P) is a validated self-report measure that is used to assess negative thinking associated with pain. The PCS-P include 13 items, which are rated on a 5-point scale ranging from 0 = "not at all true" to 4 = "very true." The items are divided across three subscales: rumination (4 items, e.g. "When my child has pain, I can't keep it out of my mind"), magnification (3 items, e.g. "When my child has pain, I keep thinking of other painful events") and helplessness (6 items, e.g. "When my child has pain, I feel like I can't go on"
Change of Parent Catastrophizing at 3 months postsurgery | 3 moths
  The Pain Catastrophizing Scale-Parent report (PCS-P) is a validated self-report measure that is used to assess negative thinking associated with pain. The PCS-P include 13 items, which are rated on a 5-point scale ranging from 0 = "not at all true" to 4 = "very true." The items are divided across three subscales: rumination (4 items, e.g. "When my child has pain, I can't keep it out of my mind"), magnification (3 items, e.g. "When my child has pain, I keep thinking of other painful events") and helplessness (6 items, e.g. "When my child has pain, I feel like I can't go on"
Change of Parent Catastrophizing at 6 months postsurgery | 6 moths
  The Pain Catastrophizing Scale-Parent report (PCS-P) is a validated self-report measure that is used to assess negative thinking associated with pain. The PCS-P include 13 items, which are rated on a 5-point scale ranging from 0 = "not at all true" to 4 = "very true." The items are divided across three subscales: rumination (4 items, e.g. "When my child has pain, I can't keep it out of my mind"), magnification (3 items, e.g. "When my child has pain, I keep thinking of other painful events") and helplessness (6 items, e.g. "When my child has pain, I feel like I can't go on"
Baseline Parent Fear of pain | 1 day presurgery
  Assess by The Fear of Pain Questionnaire-Parents (FOPQ-P): Is a validated self-report measure that used to asses fear of pain in parents with his children are in pain. The FOPQ-P include 24 ítems, which are rated on a 5-point scale ranging 0=" not at all" 5="very true". The items are divided across three subscales: fear of pain, avoidance of activities and school avoidance.
Change of Parent Fear of pain at 3 moths postsurgery | 3 moths
  Assess by The Fear of Pain Questionnaire-Parents (FOPQ-P): Is a validated self-report measure that used to asses fear of pain in parents with his children are in pain. The FOPQ-P include 24 ítems, which are rated on a 5-point scale ranging 0=" not at all" 5="very true". The items are divided across three subscales: fear of pain, avoidance of activities and school avoidance.
Change of Parent Fear of pain at 6 moths postsurgery | 6 moths
  Assess by The Fear of Pain Questionnaire-Parents (FOPQ-P): Is a validated self-report measure that used to asses fear of pain in parents with his children are in pain. The FOPQ-P include 24 ítems, which are rated on a 5-point scale ranging 0=" not at all" 5="very true". The items are divided across three subscales: fear of pain, avoidance of activities and school avoidance.
Baseline Parent Kinesiophobia | 1 day presurgery
  Assess by The Tampa Scale Kinesiophobia (TSK-11). Is a 11-item scale that measures fear of move- ment-evoked pain and injury. Scale items ranges from 0 (strongly disagree) to 4 (strongly agree) with 4 reversed- scored items. Total scores range from 25 to 56 with higher scores indicative of a greater fear of movement.
Change of Parent Kinesiophobia at 3 moths postsurgery | 3 moths
  Assess by The Tampa Scale Kinesiophobia (TSK-11). Is a 11-item scale that measures fear of move- ment-evoked pain and injury. Scale items ranges from 0 (strongly disagree) to 4 (strongly agree) with 4 reversed- scored items. Total scores range from 25 to 56 with higher scores indicative of a greater fear of movement.
Change of Parent Kinesiophobia at 6 moths postsurgery | Baseline, 3 moths, 6 months
  Assess by The Tampa Scale Kinesiophobia (TSK-11). Is a 11-item scale that measures fear of move- ment-evoked pain and injury. Scale items ranges from 0 (strongly disagree) to 4 (strongly agree) with 4 reversed- scored items. Total scores range from 25 to 56 with higher scores indicative of a greater fear of movement.
Baseline Health-related Quality of life in children | 1 day presurgery
  Assess by Pediatric Quality of Life version 4.0 Parent Version (PedsQL 4.0), which is a widely used measure of health-related quality of life in children. The PedsQL consists of 23-items, parent proxy-report forms of quality of life in younger children. Parent proxy reports have also been used for children in the age range from 2-18 years. The PedsQL assesses the following four domains of functioning: physical, emotional, social, and school and items are rated on a five-point Likert-type scale that ranges from 0 (never a problem) to 4 (almost always a problem). Items are converted to create a 0-100 scale, with higher scores reflecting higher quality of life.
Change of Health-related Quality of life in children at 3 moths postsurgery | 3 moths
  Assess by Pediatric Quality of Life version 4.0 Parent Version (PedsQL 4.0), which is a widely used measure of health-related quality of life in children. The PedsQL consists of 23-items, parent proxy-report forms of quality of life in younger children. Parent proxy reports have also been used for children in the age range from 2-18 years. The PedsQL assesses the following four domains of functioning: physical, emotional, social, and school and items are rated on a five-point Likert-type scale that ranges from 0 (never a problem) to 4 (almost always a problem). Items are converted to create a 0-100 scale, with higher scores reflecting higher quality of life.
Change of Health-related Quality of life in children at 6 moths postsurgery | 6 months
  Assess by Pediatric Quality of Life version 4.0 Parent Version (PedsQL 4.0), which is a widely used measure of health-related quality of life in children. The PedsQL consists of 23-items, parent proxy-report forms of quality of life in younger children. Parent proxy reports have also been used for children in the age range from 2-18 years. The PedsQL assesses the following four domains of functioning: physical, emotional, social, and school and items are rated on a five-point Likert-type scale that ranges from 0 (never a problem) to 4 (almost always a problem). Items are converted to create a 0-100 scale, with higher scores reflecting higher quality of life.
Baseline Pain intensity assess by parents | 1 day presurgery
  Asees by Parents' Postoperative Pain Measure (PPPM). The PPPM is completed by parents to assess children's pain following surgery and is the only validated measure of parent-report postoperative pain severity in children. Parents are asked to indicate the presence or absence of each of 15 behavioral indicators of pain.
Change of Pain intensity assess by parents at 3 moths postsurgery | 3 moths
  Asees by Parents' Postoperative Pain Measure (PPPM). The PPPM is completed by parents to assess children's pain following surgery and is the only validated measure of parent-report postoperative pain severity in children. Parents are asked to indicate the presence or absence of each of 15 behavioral indicators of pain.
Change of Pain intensity assess by parents at 6 moths postsurgery | 6 months
  Asees by Parents' Postoperative Pain Measure (PPPM). The PPPM is completed by parents to assess children's pain following surgery and is the only validated measure of parent-report postoperative pain severity in children. Parents are asked to indicate the presence or absence of each of 15 behavioral indicators of pain.

OTHER OUTCOMES:
Age | 1 day presurgery
  Age
Sex | 1 day presurgery
  Sex
Weight | 1 day presurgery
  Weight
Level of education | 1 day presurgery
  Child level of education
Situation of dependence | 1 day presurgery
  Child aid to dependency.
Socioeconomic level | 1 day presurgery
  Parents socioeconomic level

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nurse, Physiotherapy and Podiatry. University Complutense of Madrid, Madrid, Spain

REFERENCES:
- [Result] Huguet A, Miro J. The severity of chronic pediatric pain: an epidemiological study. J Pain. 2008 Mar;9(3):226-36. doi: 10.1016/j.jpain.2007.10.015. Epub 2007 Dec 21. PMID 18088558
- [Result] Miro J, Huguet A, Nieto R. Predictive factors of chronic pediatric pain and disability: a Delphi poll. J Pain. 2007 Oct;8(10):774-92. doi: 10.1016/j.jpain.2007.04.009. Epub 2007 Jul 12. PMID 17627893
- [Result] Cai Y, Lopata L, Roh A, Huang M, Monteleone MA, Wang S, Sun LS. Factors influencing postoperative pain following discharge in pediatric ambulatory surgery patients. J Clin Anesth. 2017 Jun;39:100-104. doi: 10.1016/j.jclinane.2017.03.033. Epub 2017 Apr 1. PMID 28494878
- [Result] Taylor EM, Boyer K, Campbell FA. Pain in hospitalized children: a prospective cross-sectional survey of pain prevalence, intensity, assessment and management in a Canadian pediatric teaching hospital. Pain Res Manag. 2008 Jan-Feb;13(1):25-32. doi: 10.1155/2008/478102. PMID 18301813
- [Result] Nugraha B, Gutenbrunner C, Barke A, Karst M, Schiller J, Schafer P, Falter S, Korwisi B, Rief W, Treede RD; IASP Taskforce for the Classification of Chronic Pain. The IASP classification of chronic pain for ICD-11: functioning properties of chronic pain. Pain. 2019 Jan;160(1):88-94. doi: 10.1097/j.pain.0000000000001433. PMID 30586076
- [Result] Rosenberg RE, Clark RA, Chibbaro P, Hambrick HR, Bruzzese JM, Feudtner C, Mendelsohn A. Factors Predicting Parent Anxiety Around Infant and Toddler Postoperative and Pain. Hosp Pediatr. 2017 Jun;7(6):313-319. doi: 10.1542/hpeds.2016-0166. Epub 2017 May 16. PMID 28512138
- [Result] Rabbitts JA, Fisher E, Rosenbloom BN, Palermo TM. Prevalence and Predictors of Chronic Postsurgical Pain in Children: A Systematic Review and Meta-Analysis. J Pain. 2017 Jun;18(6):605-614. doi: 10.1016/j.jpain.2017.03.007. Epub 2017 Mar 29. PMID 28363861
- [Result] Voepel-Lewis T, Caird MS, Tait AR, Farley FA, Li Y, Malviya S, Hassett A, Weber M, Currier E, de Sibour T, Clauw DJ. A cluster of high psychological and somatic symptoms in children with idiopathic scoliosis predicts persistent pain and analgesic use 1 year after spine fusion. Paediatr Anaesth. 2018 Oct;28(10):873-880. doi: 10.1111/pan.13467. PMID 30302887
- [Result] Rosenbloom BN, Page MG, Isaac L, Campbell F, Stinson JN, Wright JG, Katz J. Pediatric Chronic Postsurgical Pain And Functional Disability: A Prospective Study Of Risk Factors Up To One Year After Major Surgery. J Pain Res. 2019 Nov 12;12:3079-3098. doi: 10.2147/JPR.S210594. eCollection 2019. PMID 31814752
- [Derived] Ceniza-Bordallo G, Gomez Fraile A, Martin-Casas P, Rabbitts JA, Li R, Palermo TM, Lopez-de-Uralde-Villanueva I. Prevalence, pain trajectories, and presurgical predictors for chronic postsurgical pain in a pediatric sample in Spain with a 24-month follow-up. Pain. 2025 Jan 1;166(1):112-122. doi: 10.1097/j.pain.0000000000003330. Epub 2024 Jul 10. PMID 39047258

DOCUMENTS (3):
  • Study Protocol (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT04735211/Prot_002.pdf
  • Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT04735211/SAP_000.pdf
  • Informed Consent Form (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT04735211/ICF_001.pdf